CLINICAL TRIAL: NCT00160875
Title: A Phase II Study to Assess the Efficacy of Combined Pre-operative Chemo (CPT11, Cisplatin), Radiotherapy (External Beam, Brachytherapy), Plus Surgery for Potentially Resectable Thoracic Esophageal Cancer
Brief Title: Pre-operative Chemo (CPT11, Cisplatin), Radiotherapy, Plus Surgery for Resectable Esophageal Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-0484-C
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Cancer
Keywords: esophageal; esophagus; irinotecan; CPT11; cisplatin
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin, Irinotecan (Experimental)
  Interventions: Drug: Irinotecan hydrochloride trihydrate; Drug: Cisplatin

INTERVENTIONS:
Drug: Irinotecan hydrochloride trihydrate — Irinotecan (65mg/m2) weeks 1-2, 4-5, 7-8
Drug: Cisplatin — Cisplatin (30 mg/m2) weeks 1-2, 4-5, 7-8

SUMMARY:
Cancer of the esophagus is a very serious cancer. Studies have shown that using chemotherapy and radiation before surgery is the most promising treatment approach, with one quarter to one half of tumors shrinking by 50% or more in size after chemotherapy and radiation. In patients who have a very good response to this treatment, survival following esophagectomy has increased, although the amount of increase has varied quite a bit between the different studies. Older studies have used the drugs Cisplatin and 5-fluoruracil. Although this combination of drugs has been beneficial, we wish to use a newer combination of drugs which may be more effective for esophageal cancer. The chemotherapy drugs used in this study are Cisplatin and Irinotecan. We also want to find out what side effects these drugs cause when given with radiation, and how often these side effects occur.

DETAILED DESCRIPTION:
Historical surgical series have reported that the chance of cure with surgery alone is approximately one in four. Many phase II studies and some phase III studies have examined the role of induction (preoperative) chemotherapy and radiation. In general, these studies have demonstrated a trend to improved survival using an induction regimen with one phase III study reporting a significant improvement in survival. Two meta-analyses have failed to demonstrate a clear advantage of an induction regimen.

When these trials are reviewed, it is apparent that there is a subgroup of patients who are found at the time of resection to have had a complete pathological response to their treatment, and these patients clearly experience improved survival.

These previous trials have used older chemotherapy agents. Nevertheless, cisplatin remains one of the most active drugs available for treating solid tumours. Irinotecan is a newer drug that has demonstrated significant activity in colorectal cancer and more recently in esophageal cancer. A previous single institution trial of cisplatin and irinotecan in esophageal cancer demonstrated a significant response and acceptable toxicity.

By giving one cycle of chemotherapy alone first, it is expected that the dysphagia usually experienced by these patients will improve sufficiently and that nutritional support, i.e. feeding tube, will not be required (as has been demonstrated in a previous study of this drug combination). The same drugs will then be given concurrently with external beam radiation in order to take advantage of the radiosensitizing properties of both these drugs.

This will be followed by a boost dose of radiation, which will provide a total dose in the tumourcidal range. Surgery will follow the boost dose of radiation.

This study proposes to combine two drugs with demonstrated activity in esophageal cancer, cisplatin and Irinotecan, with radiation prior to surgery, with the hypothesis that these more active agents will offer better control of distant metastatic disease. Their radiosensitizing properties, when combined with radiation, will improve local control and provide an increased rate of pathological complete response in patients with surgically resectable esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous or adenocarcinoma or the esophagus >20 cm from the incisors, including GE junction tumors (unless of gastric origin). GE junction tumors are defined as tumors that have their center within 5 cm proximal and distal of the anatomical cardia
* Clinical T1 N1 M0, T2-3 N0-1 M0, T1-3 N0-1 M1a
* Performance status ECOG 0-2
* Medically fit for chemotherapy, radiation and esophagectomy
* Adequate bone marrow, hepatic and renal function as evidenced by the following:

Hematology:

Neutrophils > 1.5 x 109/L Platelets > 100 x 109/L

Hepatic function:

Total bilirubin < 1.25x ULN AST (SGOT) and ALT (SGPT) < 2.5 x ULN Alkaline phosphatase <2.5 x ULN

Renal function:

Serum creatinine < 160 umol/L or creatinine clearance > 60 ml/min (actual or calculated by the Cockcroft-Gault method as follows):

weight (kg) x (140 - age) K x serum creatinine*

* for serum creatinine in *mol/L, K=0.814 in man, K=0.96 in woman

  * No prior history of malignancy unless > 5 years disease free, or adequately treated nonmelanotic skin cancer or in situ carcinoma of the cervix
  * Tumor technically resectable (as defined in Section 5.4.3)

Exclusion Criteria:

* In situ or clinical T1N0M0
* Cervical esophageal tumors (within 20 cm of the incisors)
* Positive cytology of the pleura, peritoneum or pericardium
* Supraclavicular lymph node involvement
* Invasion of tracheobronchial tree proven by bronchoscopy including but not limited to tracheo-esophageal fistula
* Prior treatment for this malignancy except esophageal stenting
* Gilbert's disease
* Age < 18
* Participation in another concurrent clinical study involving study drug(s) or treatment with study drug within thirty days prior to the treatment on this study. Concurrent treatment with other experimental drugs or anticancer therapy
* Known hypersensitivity to either of study drugs or to any of their excipients.
* Pregnant or lactating women. Men and women of reproductive potential (and women < 12 months after menopause) may not participate unless they have agreed to use an effective contraceptive method while on study
* Known or suspected alcohol or drug abuse
* Other serious or concurrent illnesses that may interfere with subject compliance, adequate informed consent, determination of causality of adverse events and which in the judgement of the Investigator, would make the patient inappropriate for entry into the study
* Life expectancy < 3 months
* Peripheral neuropathy > Grade 2 (using CTC Version 2)
* Patients receiving phenytoin or phenobarbital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
pathological complete response | 1 day

SECONDARY OUTCOMES:
acute and late toxicities | 5 yrs
postoperative mortality | 1 month
disease free survival | 5 yrs
overall survival | 5 yrs
Quality of life (FACT-E) | 5 yrs
clinical complete response rate | 2 months
tumor microvessel density (pathological) | 1 day
perfusion CT parameters (radiological) | 2 months
PET scan parameters (radiological) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Darling E Gail, M.D., FRCSC, Principal Investigator — University Health Network, Toronto; Knox J Jennifer, MD,MSc,FRCPC, Principal Investigator — University Health Network, Toronto; Wong KS Rebecca, MSC, FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada